CLINICAL TRIAL: NCT04358926
Title: Hyperbaric Oxygen Therapy Effect in COVID-19 RCT (HBOTCOVID19)
Acronym: HBOTCOVID19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 120-20-ASF
Record Dates: First submitted 2020-04-21; First posted 2020-04-24 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2020-11

CONDITIONS: COVID-19; Desaturation of Blood
MeSH Terms: conditions — COVID-19 | interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Intervention Model Description: Randomized controlled study
Who Masked: Outcomes Assessor
Masking Description: The outcome assessors will receive anonymous blinded data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hyperbaric oxygen therapy (Active Comparator): 8 sessions in 4 days hyperbaric oxygen therapy
  Interventions: Device: Hyperbaric oxygen therapy
- Control (No Intervention): Standard of care

INTERVENTIONS:
Device: Hyperbaric oxygen therapy — 8 sessions in 4 days of breathing 100% oxygen in 2.2 ATA. Each session is 60 minutes. 1 meter/minute compression/decompression
  Arms: Hyperbaric oxygen therapy

SUMMARY:
The 2019-20 coronavirus disease, caused by COVID-19, is an ongoing pandemic.So far, no specific treatment has proven efficacy. Recent case series reported the use of Hyperbaric Oxygen Therapy (HBOT) on 5 severe COVID-19 patients who developed respiratory insufficiency. HBOT mechanisms of tissue oxygenation and anti-inflammatory effect may explain these findings.

The purpose of the current study is the evaluate the efficacy of HBOT in moderate-severe COVID-19 patients in a randomized controlled manner.

DETAILED DESCRIPTION:
The 2019-20 coronavirus disease, caused by COVID-19, is an ongoing pandemic. The outbreak started in Wuhan, Hubei province, China, in December 2019 and the World Health Organization (WHO) recognized it as a pandemic on 11 March 2020. Up to Apr 9. 2020 there are more than 2 million confirmed cases, and over 140,000 deaths. In Israel, COVID-19 was confirmed in more 12,000 cases and took the life of 140 victims. There are 323 mild admitted cases, 170 moderate admitted cases and 170 severe admitted cases (16.04.2020) .

Even though the general mortality rate is low (0.2-7%, country based), patients who develop Acute Respiratory Distress Syndrome (ARDS) have a significantly higher mortality rate, up to 61-90%. COVID-19 ARDS is different, causing a rapidly progressive disease including respiratory insufficiency and pulmonary fibrosis. The mechanism behind isn't clear yet, but evidence points to the direction of an acute cytokines storm which include: IL-2, IL-7, GCSF, InterferonGamma, TNF-alpha, Macrophage chemoattractant protein . Poor prognosis include high levels of IL-6 and Ferritin.

More than 160 clinical trials have been registered, but as of April 2020, there is no proven effective treatment.

The use of hyperbaric oxygen therapy (HBOT) includes breathing 100% oxygen in pressures higher than 1 absolute atmospheres (ATA), increasing the amount of oxygen dissolved in the plasma and the different tissues. In the last month, Chen et al. reported a case series of 5 severe COVID-19 patients treated with 3-8 HBOT sessions in addition to the standard therapy. In all cases, they reported an increase in oxygen saturation, arterial oxygen content,lactate levels reduction,fibrinogen levels decrease and increase in lymphocytes number.In addition, the patients chest CT showed improved signs. Symptomatic relief started following the 2nd session. No significant adverse events were reported.

These findings may be explained by the known physiological effects of HBOT, related to the SARS-CoV-2 virus pathogenesis:

1. Increased competitive binding of oxygen to the hemoglobin molecule - it has been postulated recently the SARS-CoV-2 bind to the heme component in the hemoglobin molecule and reduces the oxygen affinity to hemoglobin. During HBOT, the increased amount of available oxygen molecules increases the binding to the hemoglobin molecules. This has shown significant beneficial effects in cases of another competitive molecule such as carbon monoxide intoxication.
2. Tissue oxygenation - The oxygen content in the different tissues is multiplied by 25-30 times. This effect has two therapeutic aspects: First, overcoming pulmonary hypoxia (either shunt or VQ mismatch) by increasing the FiO2 significantly. By increasing the pulmonary oxygen gradient, oxygen diffusion increases and can overcome the inflammation in the alveoli and the thickened fibrosis caused by ARDS. Second, during HBOT, the amount of oxygen dissolved in the plasma becomes significant and enables tissue oxygenation without the need of red blood cells.
3. Anti inflammatory - HBOT reduces the following inflammatory cytokines both in the protein level and genes expression (mRNA): IL-2, TNF-alpha, IL-6, IL-1beta. The anti-inflammatory effect has been shown in chronic diseases as well as models of acute infection and massive hemorrhage.

The purpose of the current study is the evaluate the efficacy of HBOT in moderate-severe COVID-19 patients in a randomized controlled manner.

Protocol

Due to the national IRB requirements the protocol includes 2 phases:

The first phase includes 5 patients who following signing an informed consent will be treated with 8 sessions of HBOT , 2 sessions per day, in 4 consecutive days. During the sessions, the symptoms and vitals will be monitored. 1 day following the last session, revaluation will be performed.

The second phase will include 24 patients, who following signing an informed consent, will be randomized 2:1 to hyperbaric oxygen therapy group and standard of care control group. Following the randomization the patients will undergo baseline evaluation including symptoms, vitals, pulmonary function and blood tests The ratio of arterial oxygen partial pressure (PaO2 in mmHg) to fractional inspired oxygen at 5 days after enrollment was determined as the primary endpoint of the study. However, the ability to draw arterial blood gases with full COVID-19 protection gear was found to be challenging, more than usual inconvenient to the patients and many of the patients asked to avoid it (especially the draw of second arterial blood gas). Therefore, this endpoint was not completed and changed from the original protocol.

. The HBOT group patients will undergo 8 sessions of either hyperbaric oxygen therapy, 2 sessions per day, in 4 consecutive days. During the sessions, the symptoms and vitals will be monitored. 1 day following the last session, revaluation will be performed.

The control group will continue standard of care and undergo similar vitals and symptoms monitoring. 5 days after baseline evaluation, revaluation will be performed.

The long 30 days outcomes of both groups will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Within 7 days of patient's need of oxygen supply
* Positive SARS-CoV-2 RT-PCR
* At least one risk factor for bad prognosis of COVID-19: Moderate-severe Asthma, Diabetes mellitus, Cardiac conditions (congestive heart failure, coronary disease, cardiomyopathy, pulmonary hypertension), severe obesity (BMI>40), age>65, immunodeficiency, chronic liver disease.
* Respiratory insufficiency : Room Air SpO2 <94% or PaO2/FiO2<300mmHg
* Age>18
* Ability to sign an informed consent

Exclusion Criteria:

* HBOT contraindication: pneumothorax, pneumomediastinum, claustrophobia, ear/sinus disease which aren't allowed in HBOT, known chronic pulmonary disease: severe emphysema or known pulmonary bullae.
* Pregnancy
* Inability to sign an informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-04-30 (Actual); Primary Completion 2020-10-15 (Actual); Study Completion 2020-11-01 (Actual)

PRIMARY OUTCOMES:
SpO2 | 5 days after randomization
  Oxygen saturation measured in % by oxygen apparatus
NEWS Score | 5 days after randomization
  Early Warning Score (NEWS) calculated by the patient's vitals and condition
Inflammation level -CRP | 5 days after randomization
  blood CRP level
white blood cells number | 5 days after randomization
  white blood cells number
Cytokines - IL1 | 5 days after randomization
  blood IL1 level
Cytokines - IL2 | 5 days after randomization
  blood IL2 level
Cytokines - IL6 | 5 days after randomization
  blood IL6 level
Cytokines - IL10 | 5 days after randomization
  blood IL10 level
Cytokines - TNFalpha | 5 days after randomization
  blood TNFalpha level
Inflammation level - procalcitonin | 5 days after randomization
  blood procalcitonin level
Inflammation level - ferritin | 5 days after randomization
  blood ferritin level

SECONDARY OUTCOMES:
Symptoms level | 5 days after randomization
  Patient's reported symptoms including cough, dyspnea, etc.
Number of patients with IgM seroconversion | 5 days after randomization
  number of patients who developed SARS-CoV-2 IgM antibodies
Number of patients with IgG seroconversion | 5 days after randomization
  number of patients who developed SARS-CoV-2 IgG antibodies
FEV1/FVC | 5 days after randomization
  Pulmonary function tests performed bedside
Time to symptoms recovery | Within 30 days
  The measured time the patient suffered symptoms until complete recovery
Number of patients who required invasive ventilation | Within 30 days
  The number of patients who required invasive ventilation during the trial
Time to negative virus PCR | Within 30 days
  The measured time until the patient had two negative SARS-CoV-2 PCR
Mortality rate | Within 30 days
  The number of patients who died
Number of barotrauma events (safety) | 5 days after randomization
  The number of adverse events in each arm

CONTACTS AND LOCATIONS:
Overall Officials: Amir Hadanny, MD, Principal Investigator — Assaf-Harofeh Medical Center
Locations (1):
- Amir Hadanny, Ẕerifin, Israel

IPD SHARING:
Plan to Share IPD: Yes
Sharing upon specific requests will be considered
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Within 1 month of request
Access Criteria: Specific requests

REFERENCES:
- [Background] Goh KJ, Choong MC, Cheong EH, Kalimuddin S, Duu Wen S, Phua GC, Chan KS, Haja Mohideen S. Rapid Progression to Acute Respiratory Distress Syndrome: Review of Current Understanding of Critical Illness from Coronavirus Disease 2019 (COVID-19) Infection. Ann Acad Med Singap. 2020 Mar 16;49(3):108-118. PMID 32200400
- [Background] Mehta P, McAuley DF, Brown M, Sanchez E, Tattersall RS, Manson JJ; HLH Across Speciality Collaboration, UK. COVID-19: consider cytokine storm syndromes and immunosuppression. Lancet. 2020 Mar 28;395(10229):1033-1034. doi: 10.1016/S0140-6736(20)30628-0. Epub 2020 Mar 16. No abstract available. PMID 32192578
- [Background] Ruan Q, Yang K, Wang W, Jiang L, Song J. Clinical predictors of mortality due to COVID-19 based on an analysis of data of 150 patients from Wuhan, China. Intensive Care Med. 2020 May;46(5):846-848. doi: 10.1007/s00134-020-05991-x. Epub 2020 Mar 3. No abstract available. PMID 32125452
- [Background] Rogatsky GG, Mayevsky A. The life-saving effect of hyperbaric oxygenation during early-phase severe blunt chest injuries. Undersea Hyperb Med. 2007 Mar-Apr;34(2):75-81. PMID 17520858
- [Background] Weaver LK, Hopkins RO, Chan KJ, Churchill S, Elliott CG, Clemmer TP, Orme JF Jr, Thomas FO, Morris AH. Hyperbaric oxygen for acute carbon monoxide poisoning. N Engl J Med. 2002 Oct 3;347(14):1057-67. doi: 10.1056/NEJMoa013121. PMID 12362006